CLINICAL TRIAL: NCT02798315
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C -An Observational Study in Kuwait
Brief Title: Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-699
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2017-06

CONDITIONS: Chronic Hepatitis C
Keywords: Paritaprevir/r - Ombitasvir, ± Dasabuvir; Sustained Virological Response; Chronic Hepatitis C genotype 4; Observational Study; Chronic Hepatitis C genotype 1; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants With Hepatitis C Virus (HCV) Genotype 1 or 4: Participants with HCV genotype 1 or 4 receiving paritaprevir/r - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± RBV.
  The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
The interferon-free combination regimen of paritaprevir/r - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) for the treatment of chronic hepatitis C (CHC) has been shown to be safe and effective in randomized controlled clinical trials with strict inclusion and exclusion criteria under well controlled conditions.

This observational study is the first effectiveness research examining the ABBVIE REGIMEN ± RBV, used according to local label, under real world conditions in Kuwait in a clinical practice patient population.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced adult male or female participants with confirmed CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV according to standard of care and in line with the current local label.
* If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy).
* Participant must not be participating or intending to participate in a concurrent interventional therapeutic trial.

Exclusion Criteria:

* Participant must not be participating or attending in a concurrent interventional therapeutic trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hany Salaheldine, MD, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Hepatitis C Virus (HCV) Genotype 1 or 4: Participants with HCV genotype 1 or 4 receiving paritaprevir/r - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV).
Period: Overall Study
Arm/Group | Participants With Hepatitis C Virus (HCV) Genotype 1 or 4
Started | 40
Completed | 39
Not Completed | 1
Not completed — Failure to return | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With HCV Genotype 1 or 4: Participants with HCV genotype 1 or 4 receiving paritaprevir/r - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± RBV.
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Other (Not Specified) | 40
Patient Activation Measure 13 (PAM-13) [Median (Inter-Quartile Range); unit: units on a scale] — The PAM-13 item scale is a measure used to assess the patient knowledge, skill, and confidence for self-management. Based on responses to the 13-item measure, the score is calculated by adding up the raw scores (range of the sum: 13 - 52) and mapping up the value onto a scale of 0-100 indicating strength of agreement with the 13 items. A higher score indicates that the patient is likely to participate more actively in health care processes and takes more responsibility for his or her health. Population: Participants with a nonmissing baseline and end-of-treatment (EOT) assessment
  units on a scale
    number analyzed (Participants) | 37
    (all) | 55.0 [47.9 to 58.8]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 defined as the HCV ribonucleic acid (RNA) level less than 50 IU/mL 12 weeks after the last dose of study drug
Time Frame: 12 weeks (i.e. at least 70 days) after the last dose of study drug
Population: Core population: all participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
percentage of participants | 100 [91.0 to 100.0]

2. Secondary Outcome: Percentage of Participants With Virological Response at End of Treatment (EoT)
Description: Virological response defined as HCV RNA level less than 50 IU/mL.
Time Frame: Up to EoT, maximum of 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
percentage of participants | 100 [91.0 to 100.0]

3. Secondary Outcome: Percentage of Participants With Relapse at EoT
Description: Relapse defined as HCV RNA less than 50 IU/mL at EoT followed by HCV RNA greater than or equal to 50 IU/mL.
Time Frame: Up to EoT, maximum of 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
percentage of participants | 0

4. Secondary Outcome: Percentage of Participants With Breakthrough.
Description: Breakthrough defined as at least 1 documented HCV RNA less than 50 IU/mL followed by HCV RNA greater than or equal to 50 IU/mL during treatment.
Time Frame: Up to EoT, maximum of 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
percentage of participants | 0

5. Secondary Outcome: Percentage of Participants Meeting the SVR Non-response Categories of On-treatment Virologic Failure or Relapse
Description: On-treatment virologic failure defined as breakthrough (at least 1 documented HCV RNA less than 50 IU/mL followed by HCV RNA greater than or equal to 50 IU/mL during treatment) or failure to suppress (each measured on-treatment HCV RNA value greater than or equal to 50 IU/mL). Relapse (defined as HCV RNA <50 IU/mL at EoT or at the last on-treatment HCV RNA measurement followed by HCV RNA ≥50 IU/mL post-treatment).
Time Frame: 12 weeks (i.e. at least 70 days) after the last dose of study drug
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
percentage of participants
  On-treatment virologic failure | 0
  Relapse | 0

6. Secondary Outcome: Percentage of Participants Meeting the SVR Non-response Categories of Premature Study Drug Discontinuation or Missing SVR12 Data and/or None of the Above Criteria
Description: Premature study drug discontinuation category is defined as participants who prematurely discontinued study drug and who experienced no on-treatment virologic failure. The final SVR non-response category was defined as missing SVR12 data and/or none of the above criteria.
Time Frame: 12 weeks (i.e. at least 70 days) after the last dose of study drug
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
percentage of participants
  Premature study drug discontinuation | 0
  Missing SVR12 data / other | 0

7. Secondary Outcome: Adherence to ABBVIE Regimen: Percentage of the Direct-acting Antiviral (DAA) Dose Taken in Relation to the Target Dose of DAA
Description: Percentage of the DAA dose taken in relation to the target dose of DAA (cumulative dose taken divided by target dose in percent), presented as the number of participants taking > 95% to ≤ 105% of the target dose and those taking > 80% to ≤ 95% of the target dose.
Time Frame: Up to 48 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 39
Participants
  > 95% to ≤ 105% of target dose | 38
  > 80% to ≤ 95% of target dose | 1

8. Secondary Outcome: Adherence to RBV: Percentage of RBV Dose Taken in Relation to the Target Dose of RBV
Description: Percentage of the RBV dose taken in relation to the target dose of RBV (cumulative dose taken divided by target dose in percent), presented as the number of participants taking > 95% to ≤ 105% of the target dose and those taking > 80% to ≤ 95% of the target dose.
Time Frame: Up to 48 weeks
Population: Core population: all participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) and were prescribed RBV.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 33
Participants
  > 95% to ≤ 105% of target dose | 32
  > 80% to ≤ 95% of target dose | 1

9. Secondary Outcome: Adherence: Percentage of Planned Duration of RBV Taken by Participant
Time Frame: Up to 48 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of planned duration of RBV
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 33
percentage of planned duration of RBV | 101.0 (2.00)

10. Secondary Outcome: Change From Baseline in the PAM-13 Questionnaire
Description: The PAM-13 item scale is a measure used to assess the patient knowledge, skill, and confidence for self-management. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4). Based on responses to the 13-item measure, the score is calculated by adding up the raw scores (range of the sum: 13 - 52) and mapping up the value onto a scale of 0-100 indicating strength of agreement with the 13 items. A higher score indicates that the patient is likely to participate more actively in health care processes and takes more responsibility for his or her health.
Time Frame: Up to 48 weeks
Population: Core population: all participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) and contributed to the PAM-13.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 37
units on a scale | 7.60 [4.50 to 11.30]

11. Secondary Outcome: Patient Support Program (PSP) Questionnaire: Utilization of PSP Components
Description: Percentage of participants using each component of the PSP, including personal support, educational and information material (printed, online) and additional digital and mobile resources (web-portal, app, and reminders).
Time Frame: Up to EoT, maximum of 24 weeks
Population: Core population: all participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype) and who participated int he PSP.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 37
Participants
  Personal support | 28
  Educational/information material - printed | 24
  Educational/information material - online | 6
  Additional resources - web portal | 3
  Additional resources - app | 6
  Additional resources - reminders | 2

ADVERSE EVENTS:
Time Frame: Nonserious adverse events (AEs): up to 48 Weeks. Serious AEs were reported to AbbVie from the time the physician obtains the participant's authorization to use and disclose information until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment.
Arm/Group | Participants With HCV Genotype 1 or 4
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With HCV Genotype 1 or 4 (N=40)
Blood bilirubin increased (Investigations) | 2
Platelet count increased (Investigations) | 1
Overdose (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT02798315/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT02798315/SAP_001.pdf